CLINICAL TRIAL: NCT03953365
Title: Prevention of Incisional Hernia With Prophylactic Mesh in Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy. A Multicentre, Prospective, Randomised Controlled Trial
Brief Title: Prophylactic Mesh in Cytoreductive Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario Fundación Alcorcón (Other)
Responsible Party: Principal Investigator, Federico Ochando, MEDICAL DOCTOR, Hospital Universitario Fundación Alcorcón
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI 19/41
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Incisional Hernia
Keywords: hyperthermic intraperitoneal chemotherapy; cytoreduction surgery; prophylactic mesh
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- without mesh (No Intervention): Patients undergo to cytoreductive surgery and hyperthermic intraperitoneal chemotherapy without prophylactic mesh
- with mesh (Other): Patients undergo to cytoreductive surgery and hyperthermic intraperitoneal chemotherapy with prophylactic mesh
  Interventions: Procedure: Prophylactic Mesh

INTERVENTIONS:
Procedure: Prophylactic Mesh — Prophylactic Mesh after closure of the abdominal wall after Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy
  Arms: with mesh

SUMMARY:
Evaluate the effectiveness of mesh reinforcement in high-risk patients to prevent incisional hernia.

DETAILED DESCRIPTION:
Based on the hypothesis that oncological cytoreductive surgery plus hyperthermic intraperitoneal chemotherapy (HIPEC) is associated with an increased risk of developing Incisional Hernia in the postoperative period, with an expected incidence of 50% at 24 months, we designed a prospective, multicenter and randomized clinical study to demonstrate the utility of the meshes in the prevention of Incisional Hernia, hoping to reduce the incidence to 15% at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Completeness of cytoreduction after surgery (CC-SCORE) CC-0, CC-1

Exclusion Criteria:

* Completeness of cytoreduction after surgery (CC-SCORE) CC-2, CC-3

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Incisional Hernia | four years
  Prevention of Incisional Hernia

IPD SHARING:
Plan to Share IPD: No